CLINICAL TRIAL: NCT04622423
Title: Advanced Immune Gene and Cell Therapies for Liver Metastases
Brief Title: Advanced Therapies for Liver Metastases
Acronym: LiMeT
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Maria Chiara Bonini, Professor, IRCCS San Raffaele
Other Study IDs: LiMeT; 22737 (Other Grant/Funding Number: Italian Association for Cancer Research (AIRC), 5XMille call)
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC); Colorectal Cancer (CRC); Liver Metastasis
Keywords: Pancreatic ductal adenocarcinoma; Colorectal cancer; PDAC; CRC; Liver metastases; Tumor microenvironment; Immunosuppression; Immune therapy; Cell therapy; Gene therapy; Tumor infiltrating lymphocytes; ATMP
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Peripheral venous blood (from patients and healthy volunteers): additional volume collected during the diagnostic or perioperative routine/as a part of hematochemical follow-up tests/during blood donation drawings.
  2. Tissue specimens from liver MTS (from metastatic CRC and PDAC patients): extra material collected during fine-needle ago-biopsies or in therapeutic/palliative surgical resections.
  3. Tissue specimens from primary tumors (from non-metastatic PDAC patients and synchronous CRC MTS patients): extra material resected in therapeutic surgical resections.
  4. Portal blood (from non-metastatic PDAC patients): directly collected from venous vessels which will be subsequently cut and removed during standard surgical procedure, but that drain directly into the portal vein.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PDAC liver-MTS: Adult patients with clinical /radiological diagnosis/suspicious of PDAC metastatic to the liver, with subsequent cytological/histological confirmation (stage IV disease, AJCC) from liver resection/metastasectomy or core liver biopsy.
- CRC liver-MTS: Adult patients with histologically or cytologically confirmed diagnosis of CRC metastatic to the liver with indication to surgical resection (upfront or after neoadjuvant therapy).
- Primary non-MTS PDAC: Adult patients with clinical/radiological diagnosis of primary non-metastatic PDAC, candidates for surgical resection with radical intent of the primary tumor (upfront surgery or after neoadjuvant therapy). These patients will be monitored for early diagnosis of metachronous hepatic PDAC MTS by follow up testing.
- Healthy volunteers: Negative control for the clinical study.

SUMMARY:
Liver metastases (MTS) are the main cause of death for patients affected by colorectal carcinoma (CRC) and pancreatic ductal adenocarcinoma (PDAC), thus representing the major unmet clinical need for these malignancies.

Based on preliminary and published data, the investigators hypothesize that innovative immune, gene and cell therapy approaches might overcome the tolerogenic liver microenvironment and represent powerful therapeutic tools for liver MTS of PDAC and CRC.

The investigators have therefore planned an observational clinical study to enroll distinct cohorts of patients (i.e., metastatic CRC, metastatic and non-metastatic PDAC) and finely characterize, through integrated state-of-the-art -omics, the immune and non-immune microenvironment of their primary tumor and/or liver metastases as well as correlate changes in the activation status and phenotype of peripheral blood leukocytes. Healthy volunteers will be enrolled as negative controls.

The investigators aim at identifying: i) actionable tumor associated antigens (TAAs) and local immune suppressive and regulatory pathways; ii) biological parameters for early diagnosis of relapse; iii) the effect of therapies on the shaping of anti-tumor immune responses.

Data collected will be instrumental for the generation of novel advanced therapy medicinal products (ATMPs). Indeed, this protocol is part of a multi-partner translational program, supported by the AIRC 5 per Mille 2019 grant, focused on the development, validation and implementation for clinical testing of ATMPs to ameliorate the cure of CRC and PDAC and possibly help the study of other solid tumors.

Moreover, the systematic and long-term follow-up of enrolled patients will possibly point at early predictors of differential prognosis and patients' categories eligible for tailored therapies, including those with the novel ATMPs.

DETAILED DESCRIPTION:
Background and rationale - CRC and PDAC are the second and fourth most common cause of cancer death, respectively. Patients affected by these cancers die of liver MTS. Conventional therapies are active in either primary tumors but fail in metastatic disease. The effectiveness of immunotherapy by immune checkpoint blockade and adoptive cell therapy with tumor-specific T cells is only partial or temporary in MTS from solid tumors, because of local immunosuppressive mechanisms. This is particularly relevant for hepatic MTS, in which a natural tolerogenic milieu may further sustain immunosuppression induced by cancer cells and infiltrating immune cells, such as tumor associated macrophages (TAMs), myeloid-derived suppressor cells (MDSCs), neutrophils, and regulatory T or B cells.

In this regard, evidence suggests that progression of primary or metastatic CRC correlates with poor immune infiltration and inflammation. Moreover, our published results in primary PDAC support a correlation between tumor progression and a strong type 2 anti-inflammatory/immunosuppressive signature. Efficacy of chemotherapy is known to rely also on reactivation and/or repolarization of tumor targeting immune responses. Pre-surgical chemotherapy may induce beneficial effects and potentially targetable changes in the immune profile of CRC or PDAC MTS.

The investigators hypothesize that a combination of: i) direct cancer cell killing by adoptively transferred tumor-specific T cells and ii) indirect control of tumor progression via reprogramming of the tumor microenvironment would control hepatic MTS of CRC and PDAC.

Thus the investigators propose a thorough characterization of the metastatic milieu in these two cancer types to rationally shape, on the basis of similarities and differences, innovative ATMPs.

Experimental results obtained from biological samples will be correlated: i) with clinical data from patients at the time of enrollment and along their follow-up; and ii) for a subgroup of patients, with biochemical and immunological data from peripheral blood samples routinely collected as a part of their clinical follow-up, with the additional aim to identify novel biologic parameters and/or signatures to help the stratification of patients and the tailoring of treatments.

Objectives - The investigators want to study:

1. the tumor mutational burden and the composition of the metastatic tumor microenvironment in the liver;
2. the inhibitory pathways that constrain immunity in liver MTS;
3. the antigenic and clonal breadth of anti-tumor T cell responses;
4. the spatial-temporal variations of effector and regulatory immune cells upon therapy;
5. the characteristics of tumor cells and their microenvironment in liver MTS versus (vs) primary tumor;
6. the longitudinal variations of clinical parameters as well as blood-derived biological and immunological markers during the medical follow-up of patients.
7. Moreover, they want to collect and biobank patients'samples to support the validation and selection of the newl ATMPs developed by the other partners of the translational program.

The primary objectives will be:

1. to identify immune suppressive/exhaustion pathways
2. to develop a library of tumor-specific TCR (N≥5/tumor type) and identify new CAR targets (N≥1/tumor type) in CRC and PDAC MTS

Study design - This clinical protocol aims at deeply characterizing MTS tumor cells and their microenvironment, including possibly informative dynamic modifications from pro-tumor to anti-tumor profiles that may follow chemotherapy, which is administered pre-surgery (neo-adjuvant) to a substantial fraction of patients. PDAC and CRC MTS patients will be therefore characterized by either cross-sectional or longitudinal investigations on chemotherapy-naïve vs -treated patients.

In addition, the investigators aim at comparing hepatic MTS with primary tumor, in order to highlight dynamic qualitative modifications in cancer cells, immune infiltrates and not-immune microenvironment that could facilitate disease progression toward metastatic spread. These modifications may offer a window of opportunity for the optimal application of our ATMPs. To this purpose, primary non-metastatic PDAC patients undergoing surgical resection will be enrolled in this study and followed-up for monitoring the development of metachronous liver MTS, that, whenever possible, will be characterized and compared to their matched/not matched, previously collected, primary tumor samples. Peripheral blood samples at the time of liver MTS diagnosis will be also collected and analyzed. Also, in those CRC MTS patients undergoing synchronous resection of primary CRC and hepatic MTS, comparative analyses will be carried out on tumor from both sites, allowing intra- and inter-patient profiling of both tumor niches.

Moreover, results from multi-level research analyses will be correlated with clinical data collected from all patients at the time of enrollment in the study and during their clinical follow-up, whenever possible for up to 2 years, considering PDAC patients, and 3 years, considering CRC.

In particular, for metastatic CRC patients, the clinical follow-up will be associated with concurrent collection of blood samples at serial timepoints, that will be prospectively biobanked for further analyses aimed at: i) studying biological and immunological correlates of the patient's clinical status; ii) evaluating key discriminants previously identified in blood samples analyzed at the time of liver MTS surgery, to serve as early predictors of liver progression or recurrence and possibly as indicators for therapeutic stratification.

The investigators expect to collect tissue/blood samples and clinical data from at least:

* 200 metastatic CRC patients (either synchronous or metachronous);
* 150 non-metastatic PDAC patients;
* 75 synchronous PDAC MTS patients and about 20 metachronous PDAC MTS patients, the latter originally enrolled as primary non-metastatic patients for the longitudinal study, for a total of 95 metastatic PDAC patients;
* 30 healthy volunteers, as negative controls.

Different biological samples (peripheral blood, primary and/or metastatic tumor tissue, portal blood) will be collected, in the course of the standard diagnostic and therapeutic care of those patients, and will be in part directly analyzed and in part biobanked for further studies. In parallel, clinical data will be collected from patients at the time of enrollment in the study and, whenever possible, for a follow-up period of up to 2 years, for PDAC patients, and 3 years, for CRC patients.

The statistical analysis of collected data will be performed throughout the clinical study, starting 6 months after the enrollment of the first patient until 6 months after the end of patients' follow-up, for a total of 7 years. The study will last 7 years.

Different biological samples (peripheral blood, primary and/or metastatic tumor tissue, portal blood) will be collected, in the course of the standard diagnostic and therapeutic care of those patients, and will be in part directly analyzed and in part biobanked for further studies. In parallel, clinical data will be collected from patients since the time of enrollment in the study for a follow-up period of 2 years, for PDAC patients, and of 3 years, for CRC patients.

The statistical analysis of the collected clinical and experimental data will be carried out all along the duration of the clinical study, starting 6 months after the enrollment of the first patient until the end of patients' follow-up, for a total of 7 years. The study will last 7 years.

The research activities will be organized and integrated in 6 work packages (WPs):

1. Collection and biobanking of the material from patients with CRC and PDAC MTS to the liver and with primary non-metastatic resectable PDAC.
2. Definition of the tumor mutational burden, epigenetic and gene expression profile of the CRC and PDAC metastatic liver at bulk and at single cell level.
3. Evaluation of the molecular and cellular composition of CRC and, if possible, PDAC liver MTS by spatial transcriptomics technologies (NICHE-seq and Visium).
4. Characterization of the immune landscapes of CRC and, if possible, PDAC liver MTS by high dimensional flow cytometry.
5. Validation of the molecular results obtained in 2) and 4).
6. Definition of the antigenic landscape and TCR repertoire of CRC and PDAC liver MTS.

The results obtained by the above mentioned WPs will be crossed with clinical follow-up data and serve to calibrate the program activities focused on novel ATMPs development.

ELIGIBILITY:
Inclusion and exclusion criteria - CRC patients

Inclusion criteria:

1. Patients with histologically or cytologically confirmed diagnosis of CRC metastatic to the liver (stage IV disease, AJCC)
2. Patients with indication to surgical resection and/or chemotherapy treatment
3. Age ≥18
4. ECOG PS 0-1 at enrollment
5. Written informed consent
6. Patients will be treated in IRCCS San Raffaele

Exclusion criteria:

1. Pregnancy or lactation
2. Inability to provide a written informed consent
3. Extraepatic disease with the exception of selected cases in which the coexistence of extrahepatic disease does not constitute an exclusion criterion for hepatic resective surgery (for example in patients with extraepatic lesions in remission or in any case stabilized by chemotherapy)
4. Severe comorbidities (e.g. cardiac diseases, history of psychiatric disabilities, HIV, autoimmune disorders)
5. Concurrent or previous other malignancy within 5 years of study entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, or other noninvasive or indolent malignancy
6. Other conditions (medical or psychiatric) that in the judgment of Investigators would make the patient an inappropriate candidate for the study

Inclusion and exclusion criteria - PDAC patients

Inclusion criteria:

1. Patients with clinical/radiological diagnosis/suspicious of pancreatic adenocarcinoma metastatic to the liver, with subsequent cytological/histological confirmation (stage IV disease, AJCC)
2. Age ≥18
3. Karnofsky performance status ≥50
4. Metastatic pancreatic adenocarcinoma patients with histological specimens from whole liver metastasis biopsy or core liver biopsy collected at IRCCS San Raffaele and stored in the institutional biobank Centro Risorse Biologiche (CRB-OSR)
5. Written Informed consent
6. Patients with clinical/radiological diagnosis of not metastatic primary PDAC that will undergo pancreatic resection at IRCCS San Raffaele

Exclusion criteria:

1. Severe comorbidities (e.g., cardiac diseases, history of psychiatric disabilities) representing an absolute contraindication for whole or core liver metastasis biopsy
2. Pregnancy or lactation
3. Inability to provide a written informed consent
4. Metastatic pancreatic adenocarcinoma patients enrolled in other research trials entailing the analysis of the liver metastasis histological sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CRC and PDAC patients with hepatic MTS, primary non-metastatic PDAC patients and healthy volunteers. Eligible patients, chosen among those who receive health care assistance/treatment for their disease at IRCCS San Raffaele, will be asked to signing of the predisposed informed consent form in case they decide to participate in this study.
Sampling Method: Probability Sample
Enrollment: 475 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Definition of tumor mutational burden, epigenetic and gene expression profile of the CRC and PDAC metastatic liver at bulk and at single cell level | After liver metastasis/primary tumor resection/biopsy, usually within 12 months
  CRC/PDAC MTS samples will be analyzed by:
  * Whole exome DNA sequencing
  * RNA sequencing
  * ATAC sequencing
  * Single cell RNA sequencing on sorted myelomonocytic and T cells infiltrating CRC/PDAC MTS samples.
  Naive vs chemotherapy treated lesions as well as primary vs MTS lesions will be compared to evaluate chemotherapy-induced modifications and the molecular evolution in the distinct tumor sites, respectively.
Characterization of the immune landscapes of CRC and, if possible, PDAC liver MTS by high dimensional flow cytometry | For tissue specimens: immediately after tumor tissue resection/biopsy (analyses on fresh samples); for blood specimens: after blood drawing, usually within 12 months (analyses on fresh and/or thawed samples)
  Single cell suspension of CRC and PDAC MTS and paired autologous PBMCs and portal blood harvested before and after pre-operatory chemotherapy, will be analyzed by a series of parallel polychromatic high dimensional 28 color flow cytometry panels to study:
  * Conventional MHC-restricted Tab cells, the main anti-tumor effectors;
  * Innate-like T cells;
  * B cells;
  * Myelomonocytic populations involved in the stimulation or suppression of anti-tumor responses.
  Whenever available, matched primary vs MTS lesions will be compared to evaluate the immune landscapes in the distinct tumor sites.
Histological validation of the molecular results obtained in 1. and 2. | After liver metastasis/primary tumor resection/biopsy, usually within 12 months
  Validation of relevant markers and molecular pathways in terms of anatomical distribution, performed by polychromatic immunofluorence (IF, up to 6 colors) and immunohistochemistry (IHC, up to 4 colors) stainings on MTS CRC and PDAC biopsies, perilesional parenchyma and, whenever available, matched primary tumor samples. In addition to multiplex IF and IHC, some specimens will be characterized more deeply with advanced spatial proteomics technologies, such as GeoMx Digital Spatial Profiler (Nanostring).
Definition of the antigenic landscape and TCR repertoire of CRC and PDAC liver MTS | After liver metastasis/primary tumor resection/biopsy, usually within 12 months
  Identification of tumor-reactive TCRs will be pursued through different and complementary strategies:
  * The most relevant inhibitory checkpoint genes/pathways expressed by MTS-TILs will be used to enrich for tumor specificities by cell sorting harvested from CRC/PDAC MTS tumors, portal, hepatic and peripheral blood sample. After their activation, responding T cell cultures will be subject to bulk and single-cell TCR seq;
  * In samples characterized by a low percentage of MTS-TILs, single cell immune profiling will be performed in order to simultaneously determine gene expression and correctly pair chain TCR sequences from individual T cells;
  * The library of tumor-specific TCRs identified will be transiently expressed in reporter Jurkat cells to confirm their tumor antigen specificity;
  * Identification and functional validation of transmembrane molecules enriched in cancer cells as possible targets for CAR design.

SECONDARY OUTCOMES:
Evaluation of the molecular and cellular composition of CRC and, if possible, PDAC liver MTS by spatial transcriptomics technologies (NICHE-seq and Visium) | After liver metastasis/primary tumor resection/biopsy, usually within 12 months
  Application of NICHE-seq to freshly isolated human tissues using photoactivatable (cages) fluorophores able to permeate within the cells, in particular comparing ≥5 chemotherapy treated vs ≥5 naive CRC MTS samples and ≥3 PDAC MTS samples in order elucidate the high-order spatial organization of immune cell types in the NICHE-seq area and their molecular pathways, at the same time. NICHE-seq and conventional single-cell RNA seq will proceed side-by-side to compare results. Some selected specimens will be analyzed with more advanced spatial transcriptomics techniques developed in recent years, like Visium Spatial Gene Expression (10X Genomics).
Collection of clinical follow-up data | CRC patients: throughout the postoperative follow-up, for a maximum of 36 months; PDAC patients: throughout the postoperative follow-up, for a maximum of 24 months
  Overall survival (OS), disease free survival (DFS) and other follow-up parameters (patient's status, CEA levels, Ca 19-9 levels, adjuvant chemotherapy after surgery, date and site of recurrence, treatment at recurrence) will be collected and possibly correlated with the markers and pathways identified and validated in primary outcome measures.
Collection and biobanking of follow-up samples from patients with CRC and metachronous PDAC MTS to the liver | CRC: during the postoperative follow-up (up to 36 months), at six-month intervals; PDAC: during the postoperative follow-up (up to 24-months), at time of liver recurrence
  * CRC MTS patients: part of peripheral blood collected for hematochemical testing during follow-up visits
  * newly-diagnosed metachronous PDAC MTS patients, previously enrolled in the non-metastatic PDAC cohort: peripheral blood and, whenever possible, tumor tissue from liver metastasis (fine-needle bioptic sample) collected at the time of liver recurrence diagnosis, during the follow-up after the primary tumor surgery.
Biobanking of biospecimens collected from CRC and PDAC patients and from healthy donors | Throughout the protocol (7 years)
  * blood samples as detailed in the "biospecimen description" section: cryopreservation in liquid nitrogen of whole blood, plasma and purified mononuclear cells.
  * tissue samples as detailed in the "biospecimen description" section: i) formalin-fixation and paraffin embedding; ii) OCT-based embedding and cryopreservation in liquid nitrogen.
  Biobanked samples will be studied as described in 1-5, but possibly also with new state-of-the-art technologies developed in the next future.
  Moreover, they will be used to set up in vitro and in vivo systems (e.g., patient-derived organoids, tissue chips, possibly patient-derived xenograft models) to validate the efficacy and safety of the novel ATMPs developed by research program.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Bonini, MD, Principal Investigator — Vita-Salute San Raffaele University, IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lambert AW, Pattabiraman DR, Weinberg RA. Emerging Biological Principles of Metastasis. Cell. 2017 Feb 9;168(4):670-691. doi: 10.1016/j.cell.2016.11.037. PMID 28187288
- [Background] Le DT, Durham JN, Smith KN, Wang H, Bartlett BR, Aulakh LK, Lu S, Kemberling H, Wilt C, Luber BS, Wong F, Azad NS, Rucki AA, Laheru D, Donehower R, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Greten TF, Duffy AG, Ciombor KK, Eyring AD, Lam BH, Joe A, Kang SP, Holdhoff M, Danilova L, Cope L, Meyer C, Zhou S, Goldberg RM, Armstrong DK, Bever KM, Fader AN, Taube J, Housseau F, Spetzler D, Xiao N, Pardoll DM, Papadopoulos N, Kinzler KW, Eshleman JR, Vogelstein B, Anders RA, Diaz LA Jr. Mismatch repair deficiency predicts response of solid tumors to PD-1 blockade. Science. 2017 Jul 28;357(6349):409-413. doi: 10.1126/science.aan6733. Epub 2017 Jun 8. PMID 28596308
- [Background] Kitamura T, Qian BZ, Pollard JW. Immune cell promotion of metastasis. Nat Rev Immunol. 2015 Feb;15(2):73-86. doi: 10.1038/nri3789. PMID 25614318
- [Background] Zheng C, Zheng L, Yoo JK, Guo H, Zhang Y, Guo X, Kang B, Hu R, Huang JY, Zhang Q, Liu Z, Dong M, Hu X, Ouyang W, Peng J, Zhang Z. Landscape of Infiltrating T Cells in Liver Cancer Revealed by Single-Cell Sequencing. Cell. 2017 Jun 15;169(7):1342-1356.e16. doi: 10.1016/j.cell.2017.05.035. PMID 28622514
- [Background] Zitvogel L, Galluzzi L, Smyth MJ, Kroemer G. Mechanism of action of conventional and targeted anticancer therapies: reinstating immunosurveillance. Immunity. 2013 Jul 25;39(1):74-88. doi: 10.1016/j.immuni.2013.06.014. PMID 23890065
- [Background] Galon J, Costes A, Sanchez-Cabo F, Kirilovsky A, Mlecnik B, Lagorce-Pages C, Tosolini M, Camus M, Berger A, Wind P, Zinzindohoue F, Bruneval P, Cugnenc PH, Trajanoski Z, Fridman WH, Pages F. Type, density, and location of immune cells within human colorectal tumors predict clinical outcome. Science. 2006 Sep 29;313(5795):1960-4. doi: 10.1126/science.1129139. PMID 17008531
- [Background] Mlecnik B, Van den Eynde M, Bindea G, Church SE, Vasaturo A, Fredriksen T, Lafontaine L, Haicheur N, Marliot F, Debetancourt D, Pairet G, Jouret-Mourin A, Gigot JF, Hubert C, Danse E, Dragean C, Carrasco J, Humblet Y, Valge-Archer V, Berger A, Pages F, Machiels JP, Galon J. Comprehensive Intrametastatic Immune Quantification and Major Impact of Immunoscore on Survival. J Natl Cancer Inst. 2018 Jan 1;110(1). doi: 10.1093/jnci/djx123. PMID 28922789
- [Background] De Monte L, Reni M, Tassi E, Clavenna D, Papa I, Recalde H, Braga M, Di Carlo V, Doglioni C, Protti MP. Intratumor T helper type 2 cell infiltrate correlates with cancer-associated fibroblast thymic stromal lymphopoietin production and reduced survival in pancreatic cancer. J Exp Med. 2011 Mar 14;208(3):469-78. doi: 10.1084/jem.20101876. Epub 2011 Feb 21. PMID 21339327
- [Background] Galluzzi L, Buque A, Kepp O, Zitvogel L, Kroemer G. Immunological Effects of Conventional Chemotherapy and Targeted Anticancer Agents. Cancer Cell. 2015 Dec 14;28(6):690-714. doi: 10.1016/j.ccell.2015.10.012. PMID 26678337
- [Background] Nordby T, Hugenschmidt H, Fagerland MW, Ikdahl T, Buanes T, Labori KJ. Follow-up after curative surgery for pancreatic ductal adenocarcinoma: asymptomatic recurrence is associated with improved survival. Eur J Surg Oncol. 2013 Jun;39(6):559-66. doi: 10.1016/j.ejso.2013.02.020. Epub 2013 Mar 14. PMID 23498362
- [Background] Tzeng CW, Fleming JB, Lee JE, Wang X, Pisters PW, Vauthey JN, Varadhachary G, Wolff RA, Katz MH. Yield of clinical and radiographic surveillance in patients with resected pancreatic adenocarcinoma following multimodal therapy. HPB (Oxford). 2012 Jun;14(6):365-72. doi: 10.1111/j.1477-2574.2012.00445.x. Epub 2012 Feb 28. PMID 22568412
- [Background] Tjaden C, Michalski CW, Strobel O, Giese N, Hennche AK, Buchler MW, Hackert T. Clinical Impact of Structured Follow-up After Pancreatic Surgery. Pancreas. 2016 Jul;45(6):895-9. doi: 10.1097/MPA.0000000000000564. PMID 26646267
- [Background] McGranahan N, Rosenthal R, Hiley CT, Rowan AJ, Watkins TBK, Wilson GA, Birkbak NJ, Veeriah S, Van Loo P, Herrero J, Swanton C; TRACERx Consortium. Allele-Specific HLA Loss and Immune Escape in Lung Cancer Evolution. Cell. 2017 Nov 30;171(6):1259-1271.e11. doi: 10.1016/j.cell.2017.10.001. Epub 2017 Oct 26. PMID 29107330
- [Background] Fruh M, Peters S. Genomic Features of Response to Combination Immunotherapy in Lung Cancer. Cancer Cell. 2018 May 14;33(5):791-793. doi: 10.1016/j.ccell.2018.04.005. PMID 29763618
- [Background] Norelli M, Camisa B, Barbiera G, Falcone L, Purevdorj A, Genua M, Sanvito F, Ponzoni M, Doglioni C, Cristofori P, Traversari C, Bordignon C, Ciceri F, Ostuni R, Bonini C, Casucci M, Bondanza A. Monocyte-derived IL-1 and IL-6 are differentially required for cytokine-release syndrome and neurotoxicity due to CAR T cells. Nat Med. 2018 Jun;24(6):739-748. doi: 10.1038/s41591-018-0036-4. Epub 2018 May 28. PMID 29808007
- [Background] Escobar G, Barbarossa L, Barbiera G, Norelli M, Genua M, Ranghetti A, Plati T, Camisa B, Brombin C, Cittaro D, Annoni A, Bondanza A, Ostuni R, Gentner B, Naldini L. Interferon gene therapy reprograms the leukemia microenvironment inducing protective immunity to multiple tumor antigens. Nat Commun. 2018 Jul 24;9(1):2896. doi: 10.1038/s41467-018-05315-0. PMID 30042420
- [Background] Medaglia C, Giladi A, Stoler-Barak L, De Giovanni M, Salame TM, Biram A, David E, Li H, Iannacone M, Shulman Z, Amit I. Spatial reconstruction of immune niches by combining photoactivatable reporters and scRNA-seq. Science. 2017 Dec 22;358(6370):1622-1626. doi: 10.1126/science.aao4277. Epub 2017 Dec 7. PMID 29217582
- [Background] Lepore M, Mori L, De Libero G. The Conventional Nature of Non-MHC-Restricted T Cells. Front Immunol. 2018 Jun 14;9:1365. doi: 10.3389/fimmu.2018.01365. eCollection 2018. PMID 29963057
- [Background] Cortesi F, Delfanti G, Grilli A, Calcinotto A, Gorini F, Pucci F, Luciano R, Grioni M, Recchia A, Benigni F, Briganti A, Salonia A, De Palma M, Bicciato S, Doglioni C, Bellone M, Casorati G, Dellabona P. Bimodal CD40/Fas-Dependent Crosstalk between iNKT Cells and Tumor-Associated Macrophages Impairs Prostate Cancer Progression. Cell Rep. 2018 Mar 13;22(11):3006-3020. doi: 10.1016/j.celrep.2018.02.058. PMID 29539427
- [Background] Noviello M, Manfredi F, Ruggiero E, Perini T, Oliveira G, Cortesi F, De Simone P, Toffalori C, Gambacorta V, Greco R, Peccatori J, Casucci M, Casorati G, Dellabona P, Onozawa M, Teshima T, Griffioen M, Halkes CJM, Falkenburg JHF, Stolzel F, Altmann H, Bornhauser M, Waterhouse M, Zeiser R, Finke J, Cieri N, Bondanza A, Vago L, Ciceri F, Bonini C. Bone marrow central memory and memory stem T-cell exhaustion in AML patients relapsing after HSCT. Nat Commun. 2019 Mar 25;10(1):1065. doi: 10.1038/s41467-019-08871-1. PMID 30911002
- [Background] Tran E, Ahmadzadeh M, Lu YC, Gros A, Turcotte S, Robbins PF, Gartner JJ, Zheng Z, Li YF, Ray S, Wunderlich JR, Somerville RP, Rosenberg SA. Immunogenicity of somatic mutations in human gastrointestinal cancers. Science. 2015 Dec 11;350(6266):1387-90. doi: 10.1126/science.aad1253. Epub 2015 Oct 29. PMID 26516200
- [Background] Mennonna D, Maccalli C, Romano MC, Garavaglia C, Capocefalo F, Bordoni R, Severgnini M, De Bellis G, Sidney J, Sette A, Gori A, Longhi R, Braga M, Ghirardelli L, Baldari L, Orsenigo E, Albarello L, Zino E, Fleischhauer K, Mazzola G, Ferrero N, Amoroso A, Casorati G, Parmiani G, Dellabona P. T cell neoepitope discovery in colorectal cancer by high throughput profiling of somatic mutations in expressed genes. Gut. 2017 Mar;66(3):454-463. doi: 10.1136/gutjnl-2015-309453. Epub 2015 Dec 17. PMID 26681737
- [Background] Ruggiero E, Nicolay JP, Fronza R, Arens A, Paruzynski A, Nowrouzi A, Urenden G, Lulay C, Schneider S, Goerdt S, Glimm H, Krammer PH, Schmidt M, von Kalle C. High-resolution analysis of the human T-cell receptor repertoire. Nat Commun. 2015 Sep 1;6:8081. doi: 10.1038/ncomms9081. PMID 26324409
- [Background] Schumacher TN, Schreiber RD. Neoantigens in cancer immunotherapy. Science. 2015 Apr 3;348(6230):69-74. doi: 10.1126/science.aaa4971. PMID 25838375
- [Background] Balachandran VP, Luksza M, Zhao JN, Makarov V, Moral JA, Remark R, Herbst B, Askan G, Bhanot U, Senbabaoglu Y, Wells DK, Cary CIO, Grbovic-Huezo O, Attiyeh M, Medina B, Zhang J, Loo J, Saglimbeni J, Abu-Akeel M, Zappasodi R, Riaz N, Smoragiewicz M, Kelley ZL, Basturk O; Australian Pancreatic Cancer Genome Initiative; Garvan Institute of Medical Research; Prince of Wales Hospital; Royal North Shore Hospital; University of Glasgow; St Vincent's Hospital; QIMR Berghofer Medical Research Institute; University of Melbourne, Centre for Cancer Research; University of Queensland, Institute for Molecular Bioscience; Bankstown Hospital; Liverpool Hospital; Royal Prince Alfred Hospital, Chris O'Brien Lifehouse; Westmead Hospital; Fremantle Hospital; St John of God Healthcare; Royal Adelaide Hospital; Flinders Medical Centre; Envoi Pathology; Princess Alexandria Hospital; Austin Hospital; Johns Hopkins Medical Institutes; ARC-Net Centre for Applied Research on Cancer; Gonen M, Levine AJ, Allen PJ, Fearon DT, Merad M, Gnjatic S, Iacobuzio-Donahue CA, Wolchok JD, DeMatteo RP, Chan TA, Greenbaum BD, Merghoub T, Leach SD. Identification of unique neoantigen qualities in long-term survivors of pancreatic cancer. Nature. 2017 Nov 23;551(7681):512-516. doi: 10.1038/nature24462. Epub 2017 Nov 8. PMID 29132146
- [Background] Newman AM, Liu CL, Green MR, Gentles AJ, Feng W, Xu Y, Hoang CD, Diehn M, Alizadeh AA. Robust enumeration of cell subsets from tissue expression profiles. Nat Methods. 2015 May;12(5):453-7. doi: 10.1038/nmeth.3337. Epub 2015 Mar 30. PMID 25822800
- [Background] Manici S, Sturniolo T, Imro MA, Hammer J, Sinigaglia F, Noppen C, Spagnoli G, Mazzi B, Bellone M, Dellabona P, Protti MP. Melanoma cells present a MAGE-3 epitope to CD4(+) cytotoxic T cells in association with histocompatibility leukocyte antigen DR11. J Exp Med. 1999 Mar 1;189(5):871-6. doi: 10.1084/jem.189.5.871. PMID 10049951
- [Background] Tran E, Turcotte S, Gros A, Robbins PF, Lu YC, Dudley ME, Wunderlich JR, Somerville RP, Hogan K, Hinrichs CS, Parkhurst MR, Yang JC, Rosenberg SA. Cancer immunotherapy based on mutation-specific CD4+ T cells in a patient with epithelial cancer. Science. 2014 May 9;344(6184):641-5. doi: 10.1126/science.1251102. PMID 24812403
- [Background] Tran E, Robbins PF, Lu YC, Prickett TD, Gartner JJ, Jia L, Pasetto A, Zheng Z, Ray S, Groh EM, Kriley IR, Rosenberg SA. T-Cell Transfer Therapy Targeting Mutant KRAS in Cancer. N Engl J Med. 2016 Dec 8;375(23):2255-2262. doi: 10.1056/NEJMoa1609279. PMID 27959684
- [Background] Lim WA, June CH. The Principles of Engineering Immune Cells to Treat Cancer. Cell. 2017 Feb 9;168(4):724-740. doi: 10.1016/j.cell.2017.01.016. PMID 28187291

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT04622423/Prot_SAP_002.pdf